CLINICAL TRIAL: NCT04572412
Title: Low Dose Lung Radiotherapy to Treat COVID-19 Pneumonia (a Phase I Feasibility Trial)
Brief Title: Low Dose Lung Radiotherapy to Treat COVID-19 Pneumonia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lancashire Teaching Hospitals NHS Foundation Trust (Other)
Collaborators: National Institute for Health Research, United Kingdom (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 285167
Record Dates: First submitted 2020-09-29; First posted 2020-10-01 (Actual); Last update posted 2022-11-10 (Actual); Status verified 2022-11

CONDITIONS: Covid19
Keywords: SARS-CoV-2
MeSH Terms: conditions — COVID-19 | interventions — Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Low Dose Radiotherapy (Experimental): Low Dose Radiotherapy
  Interventions: Radiation: Low dose Radiotherapy

INTERVENTIONS:
Radiation: Low dose Radiotherapy — External Beam irradiation, single fraction of 0.5Gy, to be delivered within 48 hours of enrolment to study. With field to cover as close to lung edges as AP/PA technique allows.
  A further 0.5GY to the thorax given up to 96 hours apart from first fraction is permitted, if a patient had either (a) responded to the first dose but then deteriorated, however remaining better than baseline level or (b) stabilized after first dose but not fully improved.

SUMMARY:
The purpose of this study is to document the feasibility and tolerability of low dose thoracic radiotherapy in patients with WHO level 5 COVID 19 infections.

DETAILED DESCRIPTION:
Subjects will be identified following admission to hospital who test positive for COVID-19 infection. They will then be informed and consented, and eligibility confirmed and registered to study. Following this the first, sentinel patient, will be treated with 0.5Gy dose radiotherapy to cover the lungs, with heterogeneity correction. A further 0.5Gy dose can be repeated within 96 hours. There shall then be a 7 day gap prior to recruiting patient 2. The remaining patients will be recruited, treated and observed in cohorts of 3.

The patients shall then be followed up at 48 hours post Radiotherapy, 7 days post radiotherapy and 29 days post radiotherapy. With assessment of Physiological parameters, survival status, laboratory testing and imaging performed on follow up at 7 and 29 days.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 50 years.
* Patients have symptoms of COVID-19 infection as per WHO guidelines (e.g. cough, fever, dyspnea, etc.) for under 5 days from hospital admission.
* Patients are hospitalized and meet the criteria for WHO level 5 COVID pneumonia. In addition:
* SpO2 <94% on Room Air;
* Respiratory rate >20 Breaths per minute on Room Air.
* Laboratory confirmed COVID-19 infection based on PCR.
* Patients need ward-based oxygen between 28 to 40%.
* Patients able to provide witnessed verbal informed consent.
* Patient is free of other severe medical conditions that would preclude radiotherapy treatment (e.g. severe recent CVA).

Exclusion Criteria:

* Pregnant or lactating women.
* Presence of secondary infection with procalcitonin assessment at baseline.
* Patient is generating aerosols e.g. use of CPAP device.
* Hereditary syndromes known to have increase sensitivity to Radiotherapy including, but not limited to, ataxia-telangiectasia, and Njemgen Breakage Syndrome.
* History of prior thoracic radiotherapy.
* Inability to undergo radiotherapy for any reason as determined by the treating medical team.
* Alternative diagnosis for lung compromise unrelated to COVID-19 / deemed more likely than COVID-19 related lung compromise.
* Inability to consent directly.
* If patient has participated in any other COVID-19 therapy study within the last month (4 weeks).
* Pre-existing generalized pulmonary fibrosis.
* Known prior systemic use of the following drugs within the last 6 months: Bleomycin, Carmustine, Methotrexate, Busulfan, Cyclophosphamide, or Amiodarone.
* History of lung lobectomy or pneumonectomy.
* Known history of pulmonary sarcoidosis, Wegener's Granulomatosis, Systemic Lupus Erythematosus, or other autoimmune disease affecting lungs.
* Symptomatic congestive heart failure within the past 6 months including during hospitalization.
* History of recent or current malignancy receiving any cytotoxic chemotherapy or immunotherapy within the past 6 months.
* Bone marrow transplantation.
* Latent tuberculosis.
* Any solid organ transplant (renal, cardiac, liver, lung) requiring immunosuppressive therapy.
* Septic shock and organ dysfunction.
* Severe ARDS P/F ratio ≤100mmHg.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2020-11-25 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
Feasibility of Recruitment | 6 months
  Feasibility to recruit to the study.
Tolerability of Low dose Radiotherapy | 48 hours
  Proportion of patients with no decline in PaO2/FiO2 ratio (P/F Ratio) at 48 hours after each fraction of radiotherapy

SECONDARY OUTCOMES:
Withdrawal | 6 months
  The number of patients who withdraw from the study
Adverse events | 1 month
  The number of Grade 4 or higher CTCAE v5 (apart from asymptomatic lymphopenia) adverse events reported
Feasibility of biochemical analysis | 1 week
  Ability to perform lymphocyte subset, IL-6, and IL-10 analysis at baseline and 7 days post last fraction of radiotherapy

CONTACTS AND LOCATIONS:
Overall Officials: Dennis Hadjiyiannakis, Principal Investigator — LTHTR; Aashish Vyas, Principal Investigator — LTHTR
Locations (1):
- Lancashire Teaching Hospitals NHS, Preston, United Kingdom

IPD SHARING:
Plan to Share IPD: No
All data will be kept anonymized and confidential. Data will be held securely for 15 years pending further study.

REFERENCES:
- [Background] Calabrese EJ, Dhawan G. How radiotherapy was historically used to treat pneumonia: could it be useful today? Yale J Biol Med. 2013 Dec 13;86(4):555-70. PMID 24348219
- [Background] Lara PC, Burgos J, Macias D. Low dose lung radiotherapy for COVID-19 pneumonia. The rationale for a cost-effective anti-inflammatory treatment. Clin Transl Radiat Oncol. 2020 Apr 25;23:27-29. doi: 10.1016/j.ctro.2020.04.006. eCollection 2020 Jul. PMID 32373721
- [Background] Hadjiyiannakis D, Dimitroyannis D, Eastlake L, Peedell C, Tripathi L, Simcock R, Vyas A, Deutsch E, Chalmers AJ. Personal View: Low-Dose Lung Radiotherapy Should be Evaluated as a Treatment for Severe COVID-19 Lung Disease. Clin Oncol (R Coll Radiol). 2021 Jan;33(1):e64-e68. doi: 10.1016/j.clon.2020.08.003. Epub 2020 Aug 14. No abstract available. PMID 32829986
- See also: Low-Dose Whole-Lung Radiation for COVID-19 Pneumonia: Planned Day-7 Interim Analysis of a Registered Clinical Trial — https://www.medrxiv.org/content/10.1101/2020.06.03.20116988v1